CLINICAL TRIAL: NCT05711849
Title: A Phase II Randomised Sham-controlled Trial Assessing the Safety and Efficacy of Intracoronary Administration of Autologous Bone Marrow Cells in Patients With Refractory Angina
Brief Title: Assessing the Safety and Effectiveness of Intracoronary Stem Cells in Patients With Refractory Angina
Acronym: RegenCobra
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1005427
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Refractory Angina Pectoris; Refractory Angina
Keywords: Angina; Autologous stem cells; Stem cells
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Phase II randomised sham-controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Bone marrow aspiration and a single intracoronary infusion of autologous bone marrow-derived mononuclear cells.
  Interventions: Biological: Bone marrow aspiration and a single intracoronary infusion of autologous bone marrow-derived mononuclear cells.
- Sham arm (Sham Comparator): Sham bone marrow aspiration and sham cell infusion (insertion of vascular access sheath).
  Interventions: Procedure: Sham bone marrow aspiration and sham cell infusion (insertion of vascular access sheath).

INTERVENTIONS:
Biological: Bone marrow aspiration and a single intracoronary infusion of autologous bone marrow-derived mononuclear cells. — Bone marrow will be harvested from the posterior superior iliac crest under local anaesthetic, and mononuclear cells will be separated using a Ficoll technique in a certified laboratory. Later that same day, the participant will undergo an intracoronary cell infusion of the mononuclear cells. Participants will be blinded to their treatment arm (they will wear a blindfold and noise cancelling headphones for the bone marrow aspiration and cell infusion).
  Arms: Treatment arm
Procedure: Sham bone marrow aspiration and sham cell infusion (insertion of vascular access sheath). — These participants will have a sham bone marrow aspiration (a 3mm incision in the skin under local anaesthetic) and a sham intracoronary infusion procedure (the insertion of radial or femoral sheath under local anaesthetic). Participants will be blinded to their treatment arm (they will wear a blindfold and noise cancelling headphones for the sham bone marrow aspiration and sham cell infusion).
  Arms: Sham arm

SUMMARY:
REGENERATE-COBRA will examine whether autologous stem cell treatment can improve angina symptoms and quality of life for patients with refractory angina. Patients will be randomised (randomly allocated with a 50:50 chance) to either the 'treatment' or the 'sham' group - they will not know which group they are in.

In the 'treatment' group:

* Stem cells will be collected from bone marrow in the patient's hip under local anaesthetic (a bone marrow aspiration).
* Under local anaesthetic, the stem cells will be infused into the arteries that supply blood to the heart through a small tube inserted either in the wrist or the groin.
* The follow-up involves a phone call at 1 month and 12 months and clinic visit at 6 months.

In the 'sham' group:

* A sham bone marrow aspiration is performed - a 3mm nick in the skin will be made under local anaesthetic.
* A sham cell infusion is performed - a small tube is inserted either in the wrist or groin under local anaesthetic.
* The follow-up involves a phone call at 1 month and 12 months and clinic visit at 6 months.

DETAILED DESCRIPTION:
REGENERATE-COBRA is a single centre, randomised (1:1) sham-controlled clinical trial taking place at St Bartholomew's Hospital in London, UK.

* It is recruiting 110 symptomatic refractory angina patients.
* All participants will be blinded to their treatment arm. They will wear a blindfold and noise cancelling headphones for the bone marrow aspiration and the infusion procedures.
* Patients allocated to the treatment arm will undergo a bone marrow aspiration. After cell processing, the autologous bone marrow-derived mononuclear cells are infused into the coronary arteries using the stop-flow technique.
* Patients allocated to the sham arm will undergo a sham bone marrow aspiration (a 3mm nick in the skin under local anaesthetic) and a sham cell infusion (a radial or femoral sheath will be inserted under local anaesthetic).
* All patients will be followed up with a phone call at 1 month and 12 months, and a clinic visit at 6 months.
* The primary endpoint is change in Canadian Cardiovascular Society (CCS) angina score at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is older than 18 years of age
2. Symptomatic coronary artery disease (CAD) with greater than or equal to 90 days of persistent refractory angina pectoris classified as CCS Grade III or IV despite maximally tolerated guideline directed medical therapy
3. Must have attempted treatment with the maximally tolerated dose of at least two of the four approved classes of anti-anginal agents: long-acting nitrates, calcium channel blockers (either a dihydropyridine or a non-dihydropyridine), beta blockers, and ranolazine. The regimen must be stable for greater than 2 months prior to enrolment, with no intent to change the medical regimen for at least 12 months after randomisation
4. Subject has either no treatment options for revascularization by coronary artery bypass grafting or by percutaneous coronary intervention, or is otherwise unsuitable or high risk for revascularization
5. Evidence of either exercise or pharmacologically induced reversible ischemia severity by stress echo, nuclear study, PET, perfusion MRI, CT perfusion, FFRCT, FFR, iFR, or other non-hyperaemic tests.
6. Functional limitation due to refractory angina as defined by a modified Bruce exercise tolerance test duration of greater than or equal to 2 minutes but less than or equal to 8 minutes
7. Left ventricular ejection fraction (LVEF) greater than or equal to 30% within the 12- months prior to procedure (must be reassessed after any intervening myocardial infarction); the most recent LVEF assessment is used as the qualifying test
8. Subject is willing and able to sign informed consent
9. Subject is willing to comply with the specified follow-up evaluations

Exclusion Criteria:

1. Recent (within 30 days prior to enrolment) troponin or CKMB positive acute coronary syndrome (NSTEMI or STEMI).
2. Recent successful revascularization by CABG or PCI within six months prior to enrolment
3. Recent unsuccessful PCI (e.g., no relief from symptoms, failed attempt to open a chronic total occlusion) within 30 days prior to enrolment
4. The predominant manifestation of angina is dyspnoea
5. Has extra-coronary contributory causes of angina - e.g., untreated hyperthyroidism, anaemia (hgb <10 g/dL), uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg despite medications), atrial fibrillation with rapid ventricular response (consistently >100 bpm despite medications) or other tachyarrhythmia, severe aortic stenosis, hypertrophic cardiomyopathy with left ventricular outflow tract obstruction or asymmetric septal hypertrophy (concentric left ventricular hypertrophy is not an exclusion criterion), etc.
6. NYHA Class III or IV heart failure (HF), decompensated HF or hospitalisation due to HF during the 90 days prior to enrolment
7. Life threatening rhythm disorders or any rhythm disorders that would require future placement of an internal defibrillator and/or pacemaker
8. Severe chronic obstructive pulmonary disease (COPD) as indicated by a forced expiratory volume in one second (FEV1) that is less than 55% of the predicted value, or need for home daytime oxygen or oral steroids
9. Severe valvular heart disease (any valve)
10. Moderate or severe RV dysfunction by echocardiography
11. Chronic severe renal failure (estimated eGFR less than 30 mL/min/1.73m2 by the MDRD formula)
12. Any clinical condition that might interfere with the trial protocol or the subject's ability to be compliant with the trial protocol (e.g., active alcohol or drug abuse, dementia, etc.)
13. Currently enrolled in another investigational device or drug trial that has not reached its primary endpoint or that might clinically interfere with the current trial endpoints or procedures
14. Pregnant or planning pregnancy within the next 12 months (women of reproductive potential must have a negative pregnancy test within 7 days of the randomisation procedure)*
15. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.
16. Inability to tolerate dual antiplatelet therapy for 1 month if not on a chronic oral anticoagulant, or inability to tolerate a P2Y12 inhibitor for at least 1 month if on a chronic oral anticoagulant
17. Comorbidities limiting life expectancy to less than one year if recorded in patient's notes
18. Documented acute infection in patient's notes
19. Immunosuppressive medication
20. Inability to understand written and verbal English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of an intracoronary administration of autologous bone marrow-derived cells to a placebo sham treatment on Canadian Cardiovascular Society (CCS) angina scores in patients with refractory angina. | Measured pre procedure (baseline) and at 6 months post procedure
  The change in Canadian Cardiovascular Society (CCS) angina scores in all participants. Scoring is via Class I-IV where class IV is worse outcome.

SECONDARY OUTCOMES:
To compare the safety of an intracoronary administration of autologous bone marrow derived cells versus sham as measured by adverse events | Measured at 1 week post procedure, 6 months post procedure and 1 year post procedure
  Count of number of adverse events occuring in all participants
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham on myocardial ischaemic burden as measured by clinically indicated perfusion imaging | Measured pre procedure (baseline) and at 6 months post procedure
  The change in myocardial ischaemia as measured by perfusion imaging in all participants
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham on quality of life as measured by EQ-5D | Measured pre procedure (baseline) and at 6 months post procedure and 1 year post procedure
  The change in EQ-5D scores in all participants. Where the higher calculated score indicates a positive outcome.
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham on quality of life as measured by Seattle Angina Questionnaire (SAQ) | Measured pre procedure (baseline) and at 6 months post procedure and 1 year post procedure
  The change in SAQ scores in all participants. Where the higher calculated score indicates a positive outcome.
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham on total exercise time as measured by a modified Bruce protocol exercise treadmill test | Measured pre procedure (baseline) and at 6 months post procedure
  The change in total exercise time obtained by modified Bruce protocol in all participants
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham as measured by angina frequency | Measured pre procedure (baseline) and at 6 months post procedure and 1 year post procedure
  The change in number of episodes of angina occuring in a four week period prior to baseline, 6 months and 1 year visit in all participants
To compare the safety of an intracoronary administration of autologous bone marrow- derived cells versus sham as measured by major adverse cardiovascular events (MACE; defined as non-fatal stroke, non-fatal myocardial infarction and cardiovascular death) | Measured at 6 months post procedure and 1 year post procedure
  The number of major adverse events to occur measured at 6 months and 1 year in all participants
To compare the efficacy of an intracoronary administration of autologous bone marrow-derived cells versus sham as measured by change in Canadian Cardiovascular Society angina score | Measured at 6 months post procedure and 1 year post procedure
  The change in the Canadian Cardiovascular Society (CCS) angina scores in all participants. Scoring is via Class I-IV where class IV is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No